CLINICAL TRIAL: NCT03630029
Title: A Phase 1b Dose-escalating Study With RBT-1, in Healthy Volunteers and Subjects With Chronic Kidney Disease Stage 3b-4
Brief Title: RBT-1 Phase 1b Clinical Trial in Healthy Volunteers and Subjects With CKD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial has been enhanced, a new NCT(NCT03893799) listing was created.
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: REN-001
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2018-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — proto-oncogene protein c-fes-fps; tin protoporphyrin IX; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Administer a dose 12mgFeS/9mg SnPP (Other): 12 healthy volunteers will be administered a single dose of 12 mg Iron Sucrose and 9 mg of Stannous Protoporphyrin and followed for seven days.
  Interventions: Drug: FeS and SnPP
- Administer a dose 60mgFeS/45 mg SnPP (Other): 12 healthy volunteers will be administered a single dose of 60 mg of Iron Sucrose and 45 mg of Stannous Protoporphyrin and followed for seven days.
  Interventions: Drug: FeS and SnPP
- Administer a dose 120mgFeS/90mg SnPP (Other): 12 healthy volunteers will be administered a single dose of 120 mg of Iron Sucrose and 90 mg of Stannous Protoporphyrin and followed for seven days.
  Interventions: Drug: FeS and SnPP
- Administer a dose 180mgFeS/135mg SnPP (Other): 12 healthy volunteers will be administered a single dose of 180 mg and 135 mg of Stannous Protoporphyrin and followed for seven days.
  Interventions: Drug: FeS and SnPP
- Administer a dose of FeS/SnPP CKD Arm (Other): 12 subjects with stage 3 or 4 CKD will be administered a single dose of Iron Sucrose and Stannous Protoporphyrin selected from the highest dose from the prior arm that evidences the best safety profile. The subjects will be followed for seven days.
  Interventions: Drug: FeS and SnPP

INTERVENTIONS:
Drug: FeS and SnPP — Escalating doses of drug will be compared for biomarker changes
  Other Names: FeS (Iron Sucrose) SnPP (Stannous Protoporpyhrin

SUMMARY:
A Phase 1b study to evaluate the safety, tolerability and pharmacodynamic effect of RBT-1 in healthy volunteers and subjects with stage 3b-4 CKD.

DETAILED DESCRIPTION:
This is a Phase 1b, single-center, dose-escalating study to evaluate the safety, tolerability, and pharmacodynamic effect of RBT-1 in healthy volunteers and in subjects with stage 3b-4 CKD. The following biomarkers will be used as surrogate measures of protective activity: Haptoglobin, Ferritin, Bilirubin, Hemopexin, IL-10, and Heme Oxygenase-1. Additionally, the P21 biomarker will be monitored at various points of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 to 80 years (inclusive, at time of ICF).
2. Body weight <125 kg.
3. Able and willing to comply with all study procedures.
4. Female subjects must be either post-menopausal for at least 1 year or surgically sterile (tubal ligation, hysterectomy or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from Screening until 28 days after study drug administration.

   Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from screening until 28 days after study drug administration. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
5. CKD as determined by estimated glomerular filtration rate (GFR) between 15-45 ml/min as estimated using the CKD-EPI equation (CKD class 3b-4). -

Exclusion Criteria:

1. History of malignancy except carcinoma in situ in the cervix, early stage prostate cancer or non-melanoma skin cancers.
2. Use of investigational drugs or participation in another clinical trial within 30 days or 5 half-lives prior to screening, whichever is longer.
3. Serum ferritin > 500 ng/ml or who have received IV iron within 28 days of screening, or currently being treated with oral iron.
4. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
5. Regular use of drugs of abuse and/or positive findings on urinary drug screening.
6. Current tobacco use and/or positive findings on urinary cotinine screening.
7. Subjects who are severely physically or mentally incapacitated and who, in the opinion of investigator, are unable to perform the subjects' tasks associated with the protocol.
8. Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
9. Known hypersensitivity or previous anaphylaxis to RBT-1 or to components thereof. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of RBT-1 on biomarkers of cytoprotective activity | 7 days
  Measuring Haptoglobin, Ferritin, Bilirubin, Hemopexin, IL-10, and Heme Oxygenase-1, the P21 biomarker systemic levels

SECONDARY OUTCOMES:
Adverse events | 7 days
  Safety and tolerability of RBT-1 in Healthy Volunteers and subjects with CKD
Establish the optimal dose for future development | 60 days
  The highest dose of RBT-1 with the best safety and tolerability will be determined

IPD SHARING:
Plan to Share IPD: No